CLINICAL TRIAL: NCT04548609
Title: Transcranial Direct Current Stimulation (tDCS) Modulation of Neurocognitive Processes Underlying Pediatric Obsessive Compulsive Disorder (OCD)
Brief Title: Transcranial Direct Current Stimulation (tDCS) in Pediatric Obsessive Compulsive Disorder (OCD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Chief of Division of Neuropsychiatry, Director of TMS Clinic, Director of Lab for Neuropsychiatry and Neuromodulation, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020P000847
Record Dates: First submitted 2020-06-26; First posted 2020-09-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obsessive-Compulsive Disorder; Pediatric Psychiatric Disorder
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Neurodevelopmental Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Inhibitory Control/ Fear Extinction (Experimental): This arm will investigate the effect of tDCS on tasks assessing Inhibitory Control/ Fear Extinction. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation
- Inhibitory Control/ Goal-Orientated vs Habit-Based Behavior (Experimental): This arm will investigate the effect of tDCS on tasks assessing Inhibitory Control/ Goal-Orientated versus Habit-Based Behavior. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, electrodes are applied on the scalp to transmit direct current at low current amplitudes.
  Other Names: tDCS

SUMMARY:
In this study, the investigators aim to understand the role of transcranial direct current stimulation (tDCS) in modulating aberrant neurocognitive processes implicated in pediatric patients with obsessive compulsive disorder (OCD).

DETAILED DESCRIPTION:
In this study, the investigators aim to understand the role of transcranial direct current stimulation (tDCS) in modulating aberrant neurocognitive processes implicated in pediatric patients with obsessive compulsive disorder (OCD). The investigators propose two arms of the study that will investigate fear extinction learning and inhibitory control in one arm (A), and goal orientated versus habit-based behavior and inhibitory control in the other (B). All subjects will undergo three study conditions: two with active tDCS to each of two different brain targets and one under sham tDCS. The order of stimulation (sham or active tDCS) will be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient youth between the ages 10-17 years
2. Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) ≥16 (moderately severe). OCD must be determined to be the primary or co-primary diagnosis using the The Schedule for Affective Disorders and Schizophrenia for School-Age Children- Computer administered version (KSADS-COMP) based on all available information.
3. Child has a full-scale IQ≥85 as assessed on the Wechsler Abbreviated Scale of Intelligence® Second Edition (WASI®-II) (within 90% CI). To decrease participant burden, the WASI®-II will only be conducted in cases of suspected intellectual disability after meeting with the PI.
4. English speaking.

Exclusion Criteria:

1. Receiving concurrent psychotherapy for subject's OCD (except maintenance).Subjects receiving pre- established concurrent psychotherapy for at least 8 weeks regarding other psychological issues are eligible for enrollment.
2. New Treatments: Initiation of an antidepressant within 12 weeks before study enrollment or an antipsychotic 6 weeks before study enrollment. No new alternative medications, nutritional or therapeutic diets within 6 weeks of study enrolment.
3. Established Treatment changes: Any change in established psychotropic medication (e.g., antidepressants, anxiolytics, stimulant, alpha agonist) within 8 weeks before study enrollment (6 weeks for antipsychotic). Alternative medications must be stable for 6 weeks prior to baseline. Any medications must remain stable during treatment; consistent with the National Institute of Health (NIH)-funded Child Anxiety Multimodal Study (CAMS) trial, downward adjustments due to side effects may be acceptable and will be discussed with the study child and adolescent psychiatrist and the community psychiatrist.
4. Current clinically significant suicidality or individuals who have engaged in suicidal behaviors within 6 months will be excluded and referred for appropriate clinical care.
5. Meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for conduct disorder, autism, bipolar, attention deficit hyperactivity disorder (ADHD), Tourette's syndrome, schizophrenia or schizoaffective disorders
6. Youth with hoarding symptoms as they may be conceptually and genetically different from other OCD subtypes.
7. BMI less than 18.5.
8. Contraindication to tDCS: history or epilepsy, metallic implants in the head and neck, brain stimulators, vagus nerve stimulators, ventriculoperitoneal (VP) shunt, pacemakers.
9. Active substance dependence (except for tobacco).
10. Pregnant or nursing females as the effects of tDCS on pregnancy are unknown.
11. Presence of a significant and/or unstable medical illness that might lead to hospitalization during the study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Stop Signal Task | 50 minutes- 20 minutes before and immediately after a single 30 minute tDCS session
  Ability to Inhibit a Response Task
Change in Fear Extinction Recall Task | Within 12-24 hours after the tDCS session the day before
  Degree of recall to a previously extinguished conditioned stimulus
Change in Sequential Spaceship Task | 40 minutes- immediately before and 10 minutes after a 30 minute single tDCS session
  Ability to increase the proportion of Goal-Orientated versus Habit-Based Behaviour

SECONDARY OUTCOMES:
Change in EEG readings | 90 minutes- 30 minutes before and 30 minutes after a single 30 minute tDCS session
  Degree and type of change in event related potentials (ERPs) amplitudes

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD, PhD, MPH, Principal Investigator — Massachusetts General Hospital; Daniel Geller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States